CLINICAL TRIAL: NCT06545708
Title: Music and Cognitive Deficits in Self-Limited Epilepsy with Centrotemporal Spikes
Brief Title: Music Perception in SeLECTs
Acronym: EpiMUS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0084
Record Dates: First submitted 2024-07-10; First posted 2024-08-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Rolandic Epilepsy
Keywords: Epilepsy; music; childhood; neurology; rhythm; pitch; language
MeSH Terms: conditions — Epilepsy, Rolandic; Epilepsy; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: This group consists of children and adolescents between the ages of 5 and 14, diagnosed with self-limited epilepsy with centrotemporal spikes by a medical professional (epileptologist or neurologist), and in the active phase of the disorder.
  Interventions: Other: Patients
- Controls: This group consists of healthy individuals between 5 and 14 years old, with no history of epilepsy and/or other neurodevelopmental disorders.
  Interventions: Other: Patients

INTERVENTIONS:
Other: Patients — This group consists of children and adolescents between the ages of 5 and 14, diagnosed with self-limited epilepsy with centrotemporal spikes by a medical professional (epileptologist or neurologist), and in the active phase of the disorder.

SUMMARY:
Self-limited epilepsy with centrotemporal spikes (SeLECTS) is the most frequent epilepsy syndrome in children between the ages of 4 and 13 years. SeLECTS is associated in 15 to 30% of patients with specific cognitive deficits, including in particular disorders in language, visuo-spatial memory, declarative memory, and attention. SeLECTS has the potential to evolve into Landau-Kleffner syndrome, the most extreme form of SeLECTS including symptoms of auditory agnosia and aphasia, with potential risks of persistent neuropsychological impairments. In a recent study in adults who had suffered Landau-Kleffner syndrome during childhood, the investigators have shown that these patients, in addition to their known deficit in verbal short-term memory, also exhibit persistent musical difficulties during adulthood, with in particular deficit in melody and rhythm short-term memory.

In the present project, the investigators intend to enlarge the understanding of cognitive deficits generated by SeLECTS in children by investigating the integrity of music perception, both for melody and rhythm. To date, data about music perception in children with epilepsy are scarce and we do not know how distinct components of melody and rhythm perception and memory may be altered.

DETAILED DESCRIPTION:
Self-limited epilepsy with centrotemporal spikes (SeLECTS) is the most frequent epilepsy syndrome in children between the ages of 4 and 13 years. The defining electroclinical feature of SeLECTS is the presence of centrotemporal spikes on EEG between seizures. SeLECTS is associated with specific cognitive deficits in 15 to 30% of patients, including disorders in language, visuo-spatial memory, explicit memory, and attention. The centrotemporal spikes are activated in sleep and, in rare cases, the condition has the potential to evolve into an Epileptic Encephalopathy with spike- and- wave activation in sleep (EE-SWAS), including Landau-Kleffner syndrome. The latest is characterized by symptoms of auditory agnosia and aphasia, with potential risks of persistent neuropsychological impairments. In a previous study, it has been shown that these patients also exhibit persistent musical difficulties.

In the present project, the investigators intend to enlarge the understanding of cognitive deficits generated by SeLECTS in children by analyzing the integrity of music perception, both for melody and rhythm, as well as testing the potential of a musical intervention for auditory and cognitive training in children suffering from SeLECTS.

The current research plan is to explore music perception in this specific epilepsy syndrome, with behavioral testing (Experiment 1) and neuroimaging using functional Near-Infrared Spectroscopy (fNIRS) (Experiment 2), and on the long run, informed by this exploration and previous studies, the design of a musical therapeutic intervention is envisioned in order to evaluate the impact of this program on music perception, language, and memory.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged between 5 and 14 years old
* Non-opposition of parents or guardians for the child's participation in the study
* No major cognitive impairment and ability to understand and apply instructions
* Subject affiliated to a social security scheme
* Subject motivated to participate in the project
* Proficiency with the French language

For the group of control participants:

• Without neurological or psychiatric history

For the group of participants with seizure disorder:

* No neurological (except EPCT) or psychiatric history
* Diagnosis of self-limited epilepsy with centro-temporal spikes (PTSE) by a qualified healthcare professional.

Exclusion Criteria:

* Major cognitive impairment or inability to understand and apply instructions
* Individuals refusing to participate in the study
* Pregnant or breastfeeding minors

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The participants will be recruited from a population of 5 to 14 years of age. 50 healthy control participants will be recruited by posting flyers and/or by electronic message, and 50 epileptic patients will be recruited within the HFME child epileptology department (HCL). Their inclusion will be made at the CRNL or HFME by one of the study investigators.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Performance obtained in melodic tasks | 2 Years
  Comparison between controls and patients using Bayesian ANOVAs to the percentages of correct responses obtained with melodic tasks
Performance obtained in melodic tasks | 2 Years
  Comparison between controls and patients using Bayesian ANOVAs to response times obtained with melodic tasks;
Performance obtained in rhythmic tasks | 2 Years
  Comparison between controls and patients using Bayesian ANOVAs to the percentages of correct responses obtained with rhythmic tasks
Performance obtained in rhythmic tasks | 2 Years
  Comparison between controls and patients using Bayesian ANOVAs to response times obtained with rhythmic tasks.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Le Vinatier (Bât. 452),, Bron, Bron
  - Hospices Civils de Lyon, Bron, Bron

IPD SHARING:
Plan to Share IPD: No